CLINICAL TRIAL: NCT01845571
Title: Long-term Anatomic and Funcional Succes After Surgery in Eyes With Retinal Detachment
Brief Title: Retinal Detachment - Demographic and Clinical Survey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Sacu, Ass.Prof.PD.Dr., Medical University of Vienna
Other Study IDs: 13.12.2011
Record Dates: First submitted 2012-01-11; First posted 2013-05-03 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — vitreous body samples and blood plasmsa for evaluation of cytocines levels.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retinal detachment group: 400 patients patients, who received surgery due to retinal detachment exclusion: if patients had prior vitrectomy or scleral buckel if patients have no adequate follow-up

SUMMARY:
Background:

Rhegmatogenous retinal detachment is an ophthalmic emergency that, without surgical repair, often leads to blindness. The incidence is about 1/10000/year. The leading causes are myopia and aging which cause retinal tears often resulting in retinal detachment. Patients commonly experience photopsia, floaters, and peripheral visual field loss.

Two different general surgical treatment options exist for retinal detachment; scleral buckling or vitrectomy. However, the precise indications for each approach have not been well established. Correct classification of the retinal detachment is important. The first step is to decide whether an intra- or extra-ocular surgical approach is more appropriate. Simple rhegmatogenous retinal detachments are usually treated extraocularly with scleral buckling surgery, whereas more complicated cases require intraocular primary pars plana vitrectomy and one or more of gas, silicone oil, laser therapy, or cryotherapy.

Study objectives:

The purpose of this study is to evaluate different surgical techniques for the treatment of retinal detachment. Data relating to retinal status before treatment, surgical treatment, post-operative anatomy and visual acuity, post-operative OCT, and intra- and post-operative complications will be collected.

Vitreous cytokines will also be analyzed to monitor intravitreal inflammation as a result of retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

Patients who received surgery due to retinal detachment between January 2008 and Decemebr 2012.

Surgery was performed by either Ass.Prof.PD.Dr. Stefan Sacu or Prof.Dr. Michael Georgopoulos

Exclusion Criteria:

If patients had prior vitrectomy or scleral buckel. If patients had no adequate follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People will be selected from the surgery database of Ass.Prof.PD.Dr. Stefan Sacu and Prof. Dr. Michael Georgopoulos from the Medical University of Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Vision | 2 years
Aqueous cytokine Levels | baseline

SECONDARY OUTCOMES:
OCT | baseline
Surgical Data | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Sacu, Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Insitute of Ophthalmology and Optometry, Medical University of Vienna, Vienna, Austria